CLINICAL TRIAL: NCT05319080
Title: A Pilot Open-label Trial of Individualized Repetitive Transcranial Magnetic Stimulation for Patients With Auditory Verbal Hallucinations
Brief Title: Individualized Repetitive Transcranial Magnetic Stimulation for Auditory Verbal Hallucinations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator departed from institution
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Avissar, Assistant Professor of Psychiatry, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8116; K23MH119318 (NIH)
Record Dates: First submitted 2022-03-28; First posted 2022-04-08 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Hallucinations; Auditory Verbal Hallucinations
MeSH Terms: conditions — Schizophrenia; Hallucinations | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: This is an open-label study for participants with a diagnosis of either schizophrenia or schizoaffective disorder with persistent auditory verbal hallucinations (AVH) that are eligible to have repetitive transcranial magnetic stimulation (rTMS) targeting the left temporoparietal junction (TPJ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Individualized magnetic resonance imaging (MRI) guided rTMS (Experimental): Participants will receive a type of TMS called repetitive TMS (rTMS) wherein the magnetic pulses delivered will be close together in a rapid sequence. They will receive a 20-min once-daily rTMS sessions over a period of 2 weeks (weekends off), and therefore accrue a total of 10 rTMS stimulation sessions. The rTMS parameters that will be used are a frequency of 1 Hz (1 pulse per second) at an intensity of 90% of the motor threshold (MT). Therefore, the investigators will deliver 1200 continuous pulses per session/day which adds up to 12,000 pulses in total for the whole treatment.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — During the rTMS session, an electromagnetic coil is placed against the subjects scalp on the left side of the head. The electromagnet painlessly delivers a magnetic pulse that stimulates nerve cells in the region of the brain involved in speech perception.

SUMMARY:
The Repetitive Transcranial Magnetic Stimulation (rTMS) is a type of brain stimulation that uses a magnet to change activity in the brain. rTMS uses magnetic pulses to induce an electrical current in the brain to alter brain activity and function in specific areas. For example, stimulating the part of the brain controlling movement will cause parts of the foot or leg to twitch. TMS is proposed as a novel treatment for people with schizophrenia. The investigators want to see if low frequency rTMS can lessen some of the symptoms of schizophrenia, specifically auditory verbal hallucinations. Auditory verbal hallucinations describe the experience of hearing voices that are not really there.

DETAILED DESCRIPTION:
The large majority of patients with schizophrenia (Sz) experience auditory verbal hallucinations (AVH) as a core feature of their disorder. Treatment-resistant auditory verbal hallucinations (AVH) affect a third of patients with schizophrenia and can cause increased aggression, distress, suicide, and social dysfunction. The current standard of care is antipsychotic medication which can cause metabolic syndrome, sedation, orthostatic hypotension, extrapyramidal symptoms, and tardive dyskinesia among other adverse effects. Transcranial magnetic stimulation (TMS) emits a rapidly changing magnetic field over the scalp which induces current flow in underling brain tissue, either enhancing or disrupting function depending on the frequency of stimulation. It is generally well tolerated and repetitive TMS (rTMS) is currently FDA approved for treatment of depression. rTMS carries potential as an alternative treatment for schizophrenia patients with AVH who either do not respond to or do not tolerate medication. Inhibitory (1-Hz) standard TMS approaches, which use scalp-based targeting of speech perception areas such as left temporoparietal junction (TPJ) have yielded mixed results in reducing AVH, possibly due to variability of underlying brain anatomy between individual subjects. The influence of anatomical variability could be eliminated by individually positioning the TMS coil according to each patient's structural brain MRI. The proposed pilot project will investigate the clinical efficacy of open-label individualized MRI-guided TMS applied to the left TPJ in ten patients with schizophrenia or schizoaffective disorder. If the results of the pilot study show promising reductions in AVH, it will set up the foundation for a larger sham-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia or schizoaffective disorder
* Capacity and willingness to provide informed consent
* Mean Auditory Hallucination Rating Scale (AHRS) item score of greater or equal to 2
* If female and not infertile, must agree to use one of the following forms of contraception for the duration of study participation: systemic hormonal treatment, an intrauterine device (IUD) which was implanted at least 2 months prior to screening, or "double-barrier" contraception. Women of child bearing potential must have a negative pregnancy test at screening
* Right handed
* Normal hearing
* Taking an antipsychotic medication at a stable dose for at least 4 weeks. All oral and depot antipsychotics are allowable.

Exclusion Criteria:

* Substance use disorder (excluding nicotine) within last 90 days, or positive toxicology screen for any substance of abuse
* Pregnancy
* Participation in study of investigational medication/device within 4 weeks
* History of seizure, epilepsy and neurologic conditions with structural cerebral damage, including stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers, dementia, developmental disability, cerebrovascular disease, increased intracranial pressure, or central nervous system (CNS) tumors, brain surgery, head injury with loss of consciousness >1 hour or clear cognitive sequelae, intracranial metal implants, known structural brain lesion
* Subjects with devices that may be affected by TMS (pacemaker, cardioverter defibrillator, medication pump, intracardiac line, cochlear implant, implanted brain stimulator/neurostimulator)
* Subjects with suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator
* Frequent and persistent migraines
* Clinically significant skin disease
* Presence of unstable medical disorders, including those that are previously undiagnosed, untreated, inadequately treated, or active to an extent which might make participation hazardous. For example, hypertension, previous stroke, brain lesions, or heart disease
* History of prior clinically significant, adverse response to neurostimulation
* Current treatment with ototoxic medications (amino-glycosides, cisplatin)
* MRI incompatible implants
* Claustrophobia

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Avissar, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Started | 11
Completed | 5
Not Completed | 6
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5
  White | 2
  Asian | 1
  Haitian | 1
  Hispanic | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Total Number of rTMS Sessions Completed
Description: The total number of rTMS sessions completed. A session is defined as 20 minutes of rTMS. The outcome measure data comprises the cumulative count of all completed TMS sessions.
Time Frame: 2 weeks.
Population: Out of the 11 participants, 5 successfully finished all 10 treatment sessions, resulting in a combined total of 50 sessions. Additionally, two participants withdrew from the study early: one managed to complete 1 TMS treatment session, while the other completed 3 treatment sessions.
Measure: Number; unit: sessions
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 11
sessions | 54

2. Primary Outcome: Total Number of Treatment Emergent Adverse Events
Description: The total number of treatment emergent adverse events. An emergent adverse event is defined as any rTMS risk induced incident in research such as headache and seizure.
Time Frame: 2 weeks.
Population: We enrolled 11 participants in total, out of which 5 successfully completed all study procedures. Among the 6 participants who withdrew from the study midway, only 2 managed to complete a few TMS treatment sessions (the other 4 participants dropped out before the TMS treatment procedures began). As a result, we conducted an analysis in the 7 participants that completed at least one session, to assess any adverse events that occurred during the 2-week treatment session.
Measure: Number; unit: events
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 7
events | 22

3. Secondary Outcome: Change in Auditory Hallucination Rating Scale (AHRS)
Description: The AHRS is an investigator-administered scale assessing multiple characteristics of auditory verbal hallucinations. The total score ranges from 2 to 41, with higher scores indicating more severe symptoms.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 13.8 (8.8)

4. Secondary Outcome: Change in Psychotic Symptom Rating Scale (PSYRATS)- Auditory Hallucinations
Description: The PSYRATS consists of 17 items on delusions and auditory hallucinations subscales, with each item being rated from 0 (absent) to 4 (severe). The score range for the auditory hallucinations subscale is 0-44 with a higher score indicating more severe auditory hallucinations.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 12.8 (14.3)

5. Secondary Outcome: Change in Psychotic Symptom Rating Scale (PSYRATS) - Delusion Symptoms
Description: The PSYRATS consists of 17 items on delusions and auditory hallucinations, with each item being rated from 0 (absent) to 4 (severe). The score range for the delusion subscale is 0-24 with a higher score indicating more delusion symptoms.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 2 (8.7)

6. Secondary Outcome: Change in Scale for the Assessment of Positive Symptoms (SAPS)- Hallucinations
Description: The SAPS includes 34 items that focus on the positive symptoms on schizophrenia. Each item is rated on a severity scale that ranges from 0 (none) to 5 (severe). The hallucination subscale scores range from 0-35 with a higher score indicating more severe hallucinations.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 1.6 (1.3)

7. Secondary Outcome: Change in Scale for the Assessment of Positive Symptoms (SAPS)- Delusions
Description: The SAPS includes 34 items that focus on the positive symptoms on schizophrenia. Each item is rated on a severity scale that ranges from 0 (none) to 5 (severe). The delusion subscale has a range from 0-65 with a higher score indicating more severe delusion symptoms.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 0.2 (1.5)

8. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS)- General Psychopathology
Description: The PANSS rates the presence and severity of positive and negative symptoms, as well as general psychopathology associated with schizophrenia. The general psychopathology subscale is a measure of deficits in cognition with scores ranging from 16-112. Higher scores indicate more severe symptoms.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 1.8 (0.8)

9. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS)- Positive Symptoms
Description: The PANSS rates the presence and severity of positive and negative symptoms, as well as general psychopathology associated with schizophrenia. Positive symptoms defined as a symptom of schizophrenia that represents an excess or distortion of normal function, as distinct from a deficiency in or lack of normal function (compare negative symptom). Positive symptoms include delusions or hallucinations, disorganized behavior, and manifest conceptual disorganization. Positive symptom subscale ranges from 7-49 with a higher score indicating more severe symptoms.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 3.2 (4.1)

10. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS)- Negative Symptoms
Description: The PANSS rates the presence and severity of positive and negative symptoms, as well as general psychopathology associated with schizophrenia. Negative symptoms defined as a deficit in the ability to perform the normal functions of living-for example, logical thinking, self-care, social interaction, and planning, initiating, and carrying out constructive actions-as shown in apathy, blunted affect, emotional withdrawal, poor rapport, and lack of spontaneity. The negative symptoms sub scale scores range from 7-49 with a higher score indicating more severe symptoms.
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 2.4 (1.1)

11. Secondary Outcome: Change in Cardiff Anomalous Perceptions Scale (CAPS)
Description: The CAPS is a 32 item scale for measuring perceptual anomalies, that includes subscales for measuring distress, intrusiveness and frequency. A higher score indicates a higher number of perceptual anomalies, total scores range from 0 (low) to 32 (high).
Time Frame: Baseline and 4 weeks
Population: Scale scores were collected at both baseline and 4 weeks in the 5 participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 5
score on a scale | 3.6 (3.2)

12. Secondary Outcome: Number of Participants Withdrawn Resulting From a Change in Clinical Global Impression Improvement (CGI-I) Scale Score
Description: The CGI-I is a clinician-rated scale to quantify overall clinician impression of improvements in level of illness.The CGI-I is rated on a 7-point scale, to assess illness improvement. CGI-I scores range from 1 (very much improved) through to 7 (very much worse). The scale is used as a safety stop in this study. A worsening in CGI-I score of 2 or greater from baseline for two consecutive days results in withdrawal of the participant from the study.
Time Frame: Baseline and 2 weeks
Population: The investigators enrolled a total of 11 participants. Seven of 11 completed the CGI-I scale at the 2 week timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 7
Participants | 0

13. Secondary Outcome: Number of Participants Withdrawn Resulting From the Clinical Global Impression Severity (CGI-S) Scale Score
Description: The CGI-S is a clinician-rated scale to quantify overall clinician impression of illness severity. The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). The scale is used as a safety stop in this study. A score of 6 or 7 at the two week timepoint results in withdrawal of the participant from the study.
Time Frame: 2 weeks
Population: The investigators enrolled a total of 11 participants. Seven of 11 completed the CGI-I scale at the 2 week timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
Number analyzed (Participants) | 7
Participants | 0

ADVERSE EVENTS:
Time Frame: The investigators assessed participants' adverse events on a daily basis throughout the two-week TMS treatment, as well as each time participants underwent study procedures like EEG and MRI over the four-week study duration. The total time period over which adverse event data were collected was 4 weeks.
Arm/Group | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Individualized Magnetic Resonance Imaging (MRI) Guided rTMS (N=11)
Headache (Nervous system disorders) | 2
Facial pain (Nervous system disorders) | 1
Lightheadedness (Nervous system disorders) | 1
Neck discomfort (Nervous system disorders) | 1
Dizziness (Investigations) | 2
Disorientation (Investigations) | 1
Back pain (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
The study ended prematurely, resulting in a sample size that did not meet our expectations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT05319080/Prot_SAP_000.pdf